CLINICAL TRIAL: NCT02145689
Title: Long-Term Study of OnabotulinumtoxinA Treatment in Adult Patients With Upper Limb Spasticity
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn prior to enrollment due to corporate decision.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 191622-129; 2013-002327-42 (EudraCT Number)
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Muscle Spasticity; Stroke
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- onabotulinumtoxinA Dose 1 (Experimental): Up to 4 treatments of onabotulinumtoxinA Dose 1 injected into muscles of the study limb on fulfillment of the retreatment criteria.
  Interventions: Biological: onabotulinumtoxinA
- onabotulinumtoxinA Dose 2 (Experimental): Up to 4 treatments of onabotulinumtoxinA Dose 2 injected into muscles of the study limb on fulfillment of the retreatment criteria.
  Interventions: Biological: onabotulinumtoxinA

INTERVENTIONS:
Biological: onabotulinumtoxinA — Up to 4 treatments of onabotulinumtoxinA injected into muscles of the study limb on fulfillment of the retreatment criteria.
  Other Names: BOTOX®; botulinum toxin type A

SUMMARY:
This is a long-term safety and efficacy study of onabotulinumtoxinA in poststroke patients with upper limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* For patients entering from the 191622-127 study, successful completion of study 191622-127
* For patients entering directly into study 191622-129, upper limb spasticity in the elbow and shoulder due to stroke, with the most recent stroke at least 3 months ago

Exclusion Criteria:

* Spasticity in the non-study upper limb that requires treatment
* Presence of fixed contractures in of the study muscles in elbow or shoulder
* Profound atrophy of muscles to be injected
* Previous surgical intervention, nerve block, or muscle block for the treatment of spasticity in the study limb in the last 12 months
* Injection of corticosteroids or anesthetics, use of casting or dynamic splinting or constraint-induced movement therapy (CIMT) for the study limb within 3 months
* Ultrasound therapy, electrical stimulation, or acupuncture in the study limb within 1 month
* Condition other than stroke contributing to upper limb spasticity
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, and/or amyotrophic lateral sclerosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Modified Ashworth Scale-Bohannon (MAS-B) Score of Treated Muscle Groups Using a 6-Point Scale | Baseline, Up to 60 Weeks

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) of Overall Change by Physician Compared to Baseline Using a 9-Point Scale | Baseline, Up to 60 Weeks
Change from Baseline in Pain on an 11-Point Scale | Baseline, Up to 60 Weeks
Change from Baseline in the 19-Item Spasticity Impact Assessment-Upper Limb (SIA-UL) Score | Baseline, Up to 60 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan